CLINICAL TRIAL: NCT00937599
Title: The Effect of Brazil Nut Consumed on the Metabolic Profile, Oxidative Stress and Skin Microcirculatory Patterns in Obese Female Adolescents
Brief Title: Brazil Nut Consumed on the Metabolic Profile, Oxidative Stress and Nutritive Microcirculatory Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Priscila Alves Maranhão, State University of Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biovasc - 01
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Obesity
Keywords: obese; brazil nuts; oxidative stress; microcirculatory; metabolic profile
MeSH Terms: conditions — Obesity | interventions — 2S albumin, brazil nut

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Brazil Nuts (Experimental): The first group consumed the brazil nuts and the other group placebo (lactose pills)
  Interventions: Dietary Supplement: Brazil Nut

INTERVENTIONS:
Dietary Supplement: Brazil Nut — During 16 weeks the adolescents consumed 3-5 nuts/day

SUMMARY:
The purpose this research is to check if Brazil Nuts consumed improvement the metabolic profile, state redox and endothelial function in obese adolescents.

DETAILED DESCRIPTION:
The purpose this research is to check if Brazil Nuts consumed improvement the metabolic profile (lipid profile, glucose, insulin), state redox (about glutathione peroxidase, isoprostane and LDL-ox) and endothelial function (by videocapillaroscopy) in obese adolescents (12-18 years).

ELIGIBILITY:
Inclusion Criteria:

pubertal girls obese (BMI > 30 kg/m) -

Exclusion Criteria:

Consumption of nuts Loss weight before the research chronic disease (hypertension)

-

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Clinical and Experimental Research in Vascular Biology (BioVasc), Biomedical Center, State University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Maranhao PA, Kraemer-Aguiar LG, de Oliveira CL, Kuschnir MC, Vieira YR, Souza MG, Koury JC, Bouskela E. Brazil nuts intake improves lipid profile, oxidative stress and microvascular function in obese adolescents: a randomized controlled trial. Nutr Metab (Lond). 2011 May 28;8(1):32. doi: 10.1186/1743-7075-8-32. PMID 21619692